CLINICAL TRIAL: NCT02228317
Title: Emergency Medical Technician Treat-and-leave Patients Receiving Telemedicine Consultation With Emergency Medical Dispatch Physician - a Controlled Before and After Pilot-study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: Central Denmark Region (Other); Aarhus University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NRA5
Record Dates: First submitted 2014-07-11; First posted 2014-08-29 (Estimated); Last update posted 2015-12-09 (Estimated); Status verified 2014-07

CONDITIONS: Acutely Ill; Acutely Injured
Keywords: Emergency Medical Dispatch; Telemedicine; Emergency Medical Services; Pre-hospital

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Telemedicine consultation (Experimental): EMTs will systematically establish teleconsultation by either telephone or video with the EMDC-physician in all cases of non-critical illness
  Interventions: Device: Telemedicine consultation

INTERVENTIONS:
Device: Telemedicine consultation — Telemedicine consultation done by telephone or video
  Other Names: For video consultation iPAD AIR 4G/3G 16 GB will be used.; LifeSize ClearSea solution will be used for videoconferencing.; 4G/3G mobile network.; For telephone consultation Nokia C2-01 GSM telephone will be used.

SUMMARY:
A large part of acutely ill patient's access to the health care system starts by calling the emergency number 1-1-2 and thereby getting in touch with the emergency medical dispatch center (EMDC). In most cases an ambulance is dispatched and the patient is brought to the hospital. These patients are not referred by a physician (eg. a GP) and represent an unselected subpopulation of the acutely ill patients. At present, all non-critically ill patients not evaluated by a pre-hospital physician are normally be transported to hospital as category 2 (without activated emergency lightning and sirens).A part of this patient population, however, is not critically ill and a proportion of these may not need hospital admittance . Emergency medical technicians (EM) are not allowed to treat - and- leave patients without a physician's involvement. If the EMT had 24/7 online access to medical control i.e. in form of a physician present in the EMDC , the number of patients transported to hospital for assessment may be reduced as well as response times for patients actually needing ambulance transportation. This could potentially reduce the workload on the whole healthcare system involved in the management of these patients - thereby potentially reducing costs.

The objective of this study is to evaluate if a systematic telemedical assessment by an EMDC-physician of all patients who receive an ambulance but are not critically ill and would have a category 2 transport to hospital can reduce the number of the patients that are transported to hospital and save costs and time.

ELIGIBILITY:
Inclusion Criteria:

* Patients receiving an emergency ambulance after calling the EMDC Patients who are going to be admitted to a Hospital in the Central Denmark Region.
* Patients who are going to be transported as category 2 patients (non-critical illness, not requiring transport with activated lightning and sirens.

Exclusion Criteria:

* Critically ill patients (Patients who are going to be transported as category 1 patients (critical-illness, requiring immediate transport with activated sirens and warning lights )
* Patients who are not supposed to be admitted to a hospital in the Central Denmark Region

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 774 (Actual)
Dates: Start 2014-09; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Expenses related to EMDC physician vs. savings obtained by avoided admissions | Will be assessed at the time of consultation, expected to be presented within 36 months after assessment
  Cost of 24 hour EMDC physician vs. savings obtained by avoided admissions. Calculations of average transport related costs will be provided by the Prehospital Emergency Medical Services Aarhus and average cost of hospitalization for a patient hospitalized 24 hours or less at the emergency dept. will be provided by the Regional Hospital Horsens. The percentage of treat-and-leave patients in the intervention period will be compared to a historical control group represented by the average percentage of treat-and-leave patients for the previous 12 months (August 2013 to August 2014). The savings obtained by avoided admissions will be calculated by multiplying the difference in the proportion of treat and leave patients with the number of patients the previous 12 months who are receiving an ambulance after dialing 112. The EMDC physician related costs will be calculated from the present table of salary for specialist physicians in Denmark.

SECONDARY OUTCOMES:
Percentage of avoided hospital admissions | Treated-and-left or not will be assessed at the time of consultation, expected to be presented within 36 months of assessment
  Is the difference in percentage of treat-and-leave patients in the intervention period and historical control period
Response time for ambulances | Is assessed at the time the EMT registers arrival on site, expected to be presented within 36 months of assessment
  Defined as the average response time for ambulances dispatched by EMDC. The average response time is calculated as the time where the emergency medical dispatcher gets an assignment (registered manually by the dispatcher) to the arrival of the ambulance at scene (registered manually by the EMS technician). This definition of response time is predefined politically and is the gold standard for this measurement across dispatch centers in Denmark.
Hospital admission within 3 days | Will be assessed at the 72 hours after consultation, expected to be presented within 36 months of assessment
  Percentage of patients where initial hospital admission is avoided, but are admitted to hospital within 72 hours after primary contact.
Time consumption by EMDC physician | Will be assessed within 1 minute after end of consultation, expected to be presented within 36 months after assessment
  Registered as the time from receiving phone call or establishing video contact to connection is discontinued
Cause of death | Will be assessed as soon as possible after the occurence of death, normally within 24 hours, expected to be presented within 36 months of assessment
  Audit on all patients dying within 30 days of primary contact. Patient's electronic medical record will be assessed by two independent consultant physicians with no relation to EMDC in order to evaluate if death of a treat-and-leave patient can be attributed to treat-and-leave
Patient's evaluation | Will be assessed within 72 hours after end of consultation, expected to be presented within 36 months after assessment
  Patient's evaluation of prehospital care. Telephone survey of all included patients in the intervention period will be conducted within 72 hours after teleconsultation with EMDC-physician

CONTACTS AND LOCATIONS:
Locations (1):
- Prehospital Emergency Medical Services, Aarhus, Aarhus N, Denmark